CLINICAL TRIAL: NCT00943475
Title: Assessment of Hemodynamic Response and Pos-operatory Pain in Surgery of Circumcision in Children
Brief Title: Assessment of Hemodynamic Response in Surgery of Circumcision in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Marcello Fonseca Salgado Filho, Federal University of Juiz de Fora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE:0101.0.180.000-08
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-03

CONDITIONS: Children Who Need Circumcision
Keywords: DPNB, pain, hemodynamics effects, circumcision
MeSH Terms: conditions — Pain | interventions — Circumcision, Male

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anaesthesia, circumcision (Active Comparator)
  Interventions: Procedure: circumcision

INTERVENTIONS:
Procedure: circumcision — circumcision by plastbell

SUMMARY:
The surgery stress relives systemic inflammatory response by hormones and adrenergic receptors. When the pro-inflammatory mediator is higher than anti-inflammatory response, the physiologic status is impaired and the patient is more susceptible an infection and cardiovascular collapse. The anesthesia can abolish or minimize the surgery stress, improved more safety to the patient.

This study is a double blind controlled trial with 40 patients divided in two groups (EMLA and Dorsal Penile Nerve Block - DPNB) submitted a standard inhalator anesthesia and postectomy surgery by Plastbell®. The investigators will be observe heart rate, respiratory rate, arterial pressure, involuntary movements during the surgery and pain in the pos-operatory.

With this study, the investigators can define what tactic (EMLA or DPNB) associated a general anesthesia is more effective to relive the pain when children are submitted a postectomy by Plastbell®.

ELIGIBILITY:
Inclusion Criteria:

ASA status physical 1 children between 3 and 13 years old

Exclusion Criteria:

* parents don't accept the study classic circumcision

Ages: 3 Years to 13 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
local anesthesia relieve the circumcision pain | per-operatory; 1h and 24h pos-operatory

SECONDARY OUTCOMES:
local anesthesia relieve the circumcision pos-operatory pain | 1h and 24h pos-operatory

CONTACTS AND LOCATIONS:
Overall Officials: Jose murillo B Netto, Doctor, Principal Investigator — Federal University of Juiz de Fora
Locations (1):
- federal University of Juiz de Fora, Juiz de Fora, Minas Gerais, Brazil

REFERENCES:
- [Result] Serour F, Mori J, Barr J. Optimal regional anesthesia for circumcision. Anesth Analg. 1994 Jul;79(1):129-31. doi: 10.1213/00000539-199407000-00024. PMID 8010422
- [Result] Choi WY, Irwin MG, Hui TW, Lim HH, Chan KL. EMLA cream versus dorsal penile nerve block for postcircumcision analgesia in children. Anesth Analg. 2003 Feb;96(2):396-9, table of contents. doi: 10.1097/00000539-200302000-00018. PMID 12538184
- See also: Sociedade Brasileira de Anestesiologia — http://www.sba.com.br
- See also: Instituto Nacional de Cardiologia / Ministério da Saúde — http://www.inc.saude.gov.br
- See also: Society of Cardiovascular Anesthesia — http://www.scahq.org